CLINICAL TRIAL: NCT05054855
Title: Cognitive Support Technology for Postsecondary Students With Traumatic Brain Injuries (CSTPSTBI): A Randomized Clinical Trial at the Intervention Efficacy Stage of Research
Brief Title: Cognitive Support Technology for Postsecondary Students With Traumatic Brain Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-068
Record Dates: First submitted 2020-09-21; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: A minimum total of 90 students will be recruited for the study. Study personnel will recruit 30 students in each of years 2, 3, and 4. Of the 30 students per year, 15 will be randomly assigned to the full treatment intervention and 15 students will be randomly assigned to the control group. Participants will range in age from approximately 18 years to 25 years, but all ages are welcome to participate.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Treatment (Experimental): Steps of the Intervention Condition. Following an in-person session in which a pretest assessment is completed, each member of the intervention group will participate in three face-to-face sessions with the interventionist at the student's campus or at the interventionist's office to complete the CST component of the intervention.
  Interventions: Behavioral: : Cognitive Support Technology (CST)
- Abbreviated Treatment (Active Comparator): Steps of the Control Condition. Following an inperson session in which the pretest assessment is completed, each member of the control group will participate in two telephone or Skype sessions with the interventionist to discuss her or his needs for electronic cognitive supports. An abbreviated version of Scherer's (2012) MPT assessment will be administered via telephone or Skype in the first of these virtually-administered sessions. In the second telephone or Skype session, the interventionist will summarize the results of the abbreviated MPT assessment, suggest a variety of cognitive enhancement apps for tablet computers or smart phones that the control group participant can consider.
  Interventions: Behavioral: : Cognitive Support Technology (CST)

INTERVENTIONS:
Behavioral: : Cognitive Support Technology (CST) — Cognitive Support Technology (CST) products and strategies are used to help people with disabilities compensate for or accommodate cognitive limitations (including those related to interpersonal communication and social cognition) that present difficulties for them in the performance of desired social roles, especially education and employment.
  CSTs may be mainstream everyday technologies such as tablet computers or they may be specialized devices designed for specific goals such as step-by-step instruction in the performance of a particular task (Scherer, 2012).

SUMMARY:
This study will fill important knowledge gaps in the availability of best practices that use innovative methods to integrate the cognitive and vocational needs of students with TBI who will be transitioning from 2- and 4-year postsecondary education to employment. Best practices exist from the assistive technology (AT) field to help people compensate for cognitive impairments, and from the vocational rehabilitation (VR) field to enhance employment outcomes for individuals with disabilities. However, these practices have not been integrated to provide needed supports and services to improve the employment outcomes of students with TBI. The study's goal is to expand the availability of innovative practices by testing the efficacy of a technology-driven, long-term, and resource-rich individualized support program that merges assistive technology for cognition and vocational rehabilitation practices. The end products will include technology application guidelines, training and procedural manuals, and resource information that rehabilitation professionals and students with TBI can utilize to enhance technology and mentoring proficiency, academic success, self-determination, and long-term career success for students with TBI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TBI
* Enrolled in a degree program at two-year and four-year colleges or universities
* Live within a 60-mile radius of Kent, Ohio

Exclusion Criteria:

* No exclusion criteria will be applied

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Grade Point Average (GPA) | Baseline (enrollment in study) and 1 year (study completion)
  Participant GPA

SECONDARY OUTCOMES:
Change in Post-Secondary Enrollment Status | Baseline (enrollment in study) and 1 year (study completion)
  % of participants still enrolled in a postsecondary program
Change in Satisfaction with transportation access | Baseline (enrollment in study) and 1 year (study completion)
  Measured using single item 5-point Likert question on questionnaire
Change in Satisfaction with Social Support | Baseline (enrollment in study) and 1 year (study completion)
  Measured using single item 5-point Likert question on questionnaire
Change in Current Employment Status | Baseline (enrollment in study) and 1 year (study completion)
  Three items on questionnaire including dichotomous employment question (e.g., are you employed?), if yes, number of hours employed and weekly earnings.
Change in % of Participants Receiving Disability Benefits | Baseline (enrollment in study) and 1 year (study completion)
  Whether participants receive SSDI and/or SSI benefits or not
Change in Overall health status | Baseline (enrollment in study) and 1 year (study completion)
  Measured using RAND 36-item Health Survey 1.0 All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Change in Depression Symptoms | Baseline (enrollment in study) and 1 year (study completion)
  Measured using Beck Depression Inventory- II (BDI-II) The BDI-II is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3. The maximum total score is 63. A higher score indicates a higher level of depressive symptomology.
Change in Acceptance of disability | Baseline (enrollment in study) and 1 year (study completion)
  Measured using the Acceptance of Disability Scale- Short Form There are 50 self-report items. Each item, provides a single score that ranges from 1 (low acceptance of disability) to 6 (high acceptance of disability). An overall acceptance of disability score is derived by summing all items, with 300 as the highest possible score. Low acceptance scores fall below 175, whereas high acceptance scores range from 176 to 300
Change in Perceived Stress | Baseline (enrollment in study) and 1 year (study completion)
  Measured using the Perceived Stress Scale- 10. PSS-10 scores are obtained by reversing the scores on the four positive items, e.g., 0=4, 1=3, 2=2, etc. and then summing across all 10 items. Items 4,5, 7, and 8 are the positively stated items. The highest score possible is 40 while the lowest score possible is 0. Higher score indicates higher levels of perceived stress.
Change in Quality of Life (QoL) | Baseline (enrollment in study) and 1 year (study completion)
  Measured using the Quality of Life Scale There are 16 items scored on a seven-point Likert scale. The seven responses are "delighted" (7), "pleased" (6), "mostly satisfied" (5),"mixed" (4), "mostly dissatisfied" (3), "unhappy" (2),"terrible" (1).The QOLS is scored by adding up the score on each item to yield a total score for the instrument. Scores can range from 16 to 112 with higher scores representing a higher reported quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No